CLINICAL TRIAL: NCT02318823
Title: Effects of Beer (Alcohol) on Social Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKNZ 2014-369
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: social neuroscience; emotion; face recognition; empathy; beer; alcohol; social cognition
MeSH Terms: interventions — Beer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beer (alcoholic) followed by placebo (non-alcoholic) (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has two treatment conditions in the same subject.
  Interventions: Other: Beer (alcoholic); Other: Placebo (non-alcoholic beer)
- Placebo (non-acoholic beer) followed by Beer (alcoholic) (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has two treatment conditions in the same subject.
  Interventions: Other: Beer (alcoholic); Other: Placebo (non-alcoholic beer)

INTERVENTIONS:
Other: Beer (alcoholic) — Beer (individually calculated amount aiming to achieve a blood-alcohol-centration of 0.4g/kg)
Other: Placebo (non-alcoholic beer) — Non-alcoholic beer serves as Placebo.

SUMMARY:
The present study aims to evaluate effects of beer (alcohol) on social cognition.

DETAILED DESCRIPTION:
Alcohol is one of the most widely used recreational drugs and it is often used in social settings to enhance sociability. There are few data showing that acute alcohol consumption affects facial emotion recognition. However the acute effects of alcohol in social drinkers on different aspects of social cognition are largely unknown. In the present study, we will therefore evaluate effects of beer (alcohol) on social cognition. The study will include 60 subjects (30 male, 30 female) and use a placebo-controlled, crossover design with the two experimental conditions alcoholic beer (individually calculated amount aiming to achieve a blood-alcohol concentration of 0.4g/kg), and non-alcoholic beer (placebo). We primarily aim to evaluate whether beer (alcohol) affects the ability to correctly decode emotions in facial expressions using different facial emotion recognition Tasks. Additionally, appraisal of visual erotic stimuli following alcohol consumption will be evaluated. Subjective social and mood effects will be assessed using validated questionnaires. Blood samples will be collected to assess plasma levels of the "social hormone" oxytocin as well as blood alcohol levels to test possible associations with effects on emotional processing.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years
2. Sufficient understanding of the German language
3. Subjects understand the procedures and the risks associated with the study
4. Participants must be willing to adhere to the protocol and sign the consent form
5. Participants must be willing to refrain from drinking alcohol in the evening preceding the study session
6. Participants must be willing to abstain from excessive drinking and from taking illicit psychoactive drugs during the study.
7. Participants must be willing not to eat or drink xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) 3 h prior to the study session
8. Participants must be willing not to drive a traffic vehicle or to operate machines for 3h after the sessions
9. Women must have a negative pregnancy test at the beginning of each session.

Exclusion Criteria:

1. Chronic or acute medical condition.
2. Current or previous personal history of psychotic or major affective disorder.
3. Prior or current alcohol abuse, dangerous drinking behavior (>15 points in the AUDIT questionnaire).
4. Family history of alcoholism (first-degree relative).
5. Alcohol hypersensitivity
6. Prior illicit drug use (except Tetrahydrocannabinol (THC)-containing products) more than 15 times or any time within the previous week.
7. Use of medications that are contraindicated or interfere otherwise with the effects of the study (monoamine oxidase inhibitors, antidepressants, sedatives etc.)
8. Pregnant or nursing women.
9. Participation in another clinical trial (currently or within the last 30 days).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effect of beer (alcohol) on emotion recognition | 3 hours

SECONDARY OUTCOMES:
Effect of beer (alcohol) on empathy and social behavior | 3 hours
Subjective effects of beer (alcohol) | 3 hours
Effect of beer (alcohol) on appraisal of visual erotic stimuli | 3 hours
Effects of beer (alcohol) on plasma oxytocin | 3 hours
Effect modulation by genetic polymorphisms | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Dolder PC, Holze F, Liakoni E, Harder S, Schmid Y, Liechti ME. Alcohol acutely enhances decoding of positive emotions and emotional concern for positive stimuli and facilitates the viewing of sexual images. Psychopharmacology (Berl). 2017 Jan;234(1):41-51. doi: 10.1007/s00213-016-4431-6. Epub 2016 Sep 19. PMID 27640999